CLINICAL TRIAL: NCT05576311
Title: Conducting Focus Groups With Patients and Healthcare Practitioners to Inform the Development of a Sensor Which Measures Urine Flow, Volume and Voiding Patterns, in Order to Diagnose Pathologies of the Urinary System
Brief Title: Codesign of an Optical Device to Measure Urine Flow and Volume
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Teesside University (Other)
Collaborators: South Tees Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, John S. Young, Professor of Translational Healthcare, Teesside University
Other Study IDs: 10852
Record Dates: First submitted 2022-10-05; First posted 2022-10-12 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Urinary Incontinence; Urinary Retention; Urinary Tract Infections; Overactive Bladder; Benign Prostatic Hyperplasia; Underactive Bladder
MeSH Terms: conditions — Urinary Incontinence; Urinary Retention; Urinary Tract Infections; Urinary Bladder, Overactive; Prostatic Hyperplasia; Urinary Bladder, Underactive | interventions — Focus Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Focus Group — Focus Groups to capture information about the need for innovation in the diagnosis and monitoring of urinary symptoms.

SUMMARY:
The study is seeking to understand the needs of patients and healthcare practitioners for an innovation in the way that changes in bladder function are assessed. This information will be used in the design and evaluation of a device, being developed in parallel, that assesses changes to the volume and flow of urine in order to determine changes in bladder function.

In order to ensure development is optimal, the principal research objective is therefore to understand the needs of patients and healthcare practitioners (ranging from care home staff and GPs in primary care, to urologists in tertiary referral centres).

ELIGIBILITY:
Inclusion criteria The participant is willing and able to give informed consent for participation in the study.

Aged 18 years or above. Male or Female.

Exclusion criteria The participant is unwilling or unable to give informed consent for participation in the study.

Aged 17 years or younger.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be patients with urinary symptoms referred to Consultant Urological Surgeon Ms Mehwash Nadeem at the James Cook Hospital, Middlesbrough or the Friarage Hospital, Northallerton.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Understanding the needs of patients and healthcare practitioners for an innovation in the way that changes in bladder function are assessed. | November 2022 - February 2023
  For ~45 participants for each of two categories, patients and healthcare practitioners, focus groups will chart the difficulties, needs, potential solutions, and concerns of all participants, as well as collect their input on the prototype that we are developing. Their responses will be coded, grouped, and summarised, to create a set of guidelines aiding the future development of solutions for urinary disorders.

IPD SHARING:
Plan to Share IPD: No